CLINICAL TRIAL: NCT02734121
Title: Pre-consultation Educational Group Intervention to Improve Shared Decision-Making for Postmastectomy Breast Reconstruction
Brief Title: PEGI to Improve Shared Decision-Making for Breast Reconstruction
Acronym: PEGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-7227-CE
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast reconstruction; shared decision making; decision support intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational group intervention (Experimental): The pre-consultation educational group intervention will be 2 hours in duration on the morning of the consultation and will be facilitated by a dedicated social worker from psycho-oncology.
  Interventions: Behavioral: pre-consultation educational group intervention
- Standard Care (No Intervention): Routine pre-consultation education

INTERVENTIONS:
Behavioral: pre-consultation educational group intervention — Incorporates the key components of shared decision-making and decision support with the philosophy of delivering supportive care to cancer patients.
  * Surgeon (40 mins): treatment options for breast reconstruction with indications/ contraindications, advantages / disadvantages, expected post-operative course, aesthetic result and complications with probabilities
  * Registered nurse (20 mins): preparing for surgery, postoperative recovery and how to navigate the health care system
  * Social worker (30 mins): values clarification exercise
  * Breast reconstruction patient volunteers (30 mins) questions and answers about their personal experience
  Arms: Educational group intervention

SUMMARY:
The purpose of this study is to determine the effectiveness of a pre-consultation decision support workshop for breast reconstruction after breast cancer, in facilitating the decision-making process, compared to routine pre-surgical education.

DETAILED DESCRIPTION:
Postmastectomy breast reconstruction is becoming increasingly utilized in breast cancer patients to provide surgical restoration of the breast mounds. The breast reconstruction discussions can be highly complex, as there are many different techniques, timing, and complications that are unique to each procedure. However ¼ of women report being dissatisfied with some component of their cancer or reconstructive care. Failure of the physician to provide adequate information about treatment options is the most frequent source of cancer patient dissatisfaction and breast reconstruction patients have expressed a need for further information regarding the complex decision to pursue breast reconstruction. In such scenarios of complex medical decision-making, decision support techniques may be an effective solution to information provision and shared decision-making. As a result, the investigators developed a pre-consultation educational group intervention delivered in a group setting for women considering breast reconstruction, with the aims to fill an existing information-gap, promote high-quality decision-making and enhance decision self-efficacy and other decision measures. This study will evaluate the educational group intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age.
2. Seeking consultation for delayed Post Mastectomy Breast Reconstruction, or prophylactic mastectomy and immediate Post Mastectomy Breast Reconstruction for breast cancer prevention.

Exclusion Criteria:

1. Chest wall or atypical breast malignancy that require chest wall reconstruction.
2. Active invasive or in situ breast cancer.
3. Consultation for breast revision or nipple reconstruction only.
4. Patient cannot read or write in English.
5. Cognitive impairment or uncontrolled psychiatric diagnosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | Change from baseline decision conflict at 1 week after surgical consultation
  Decision conflict scale measures personal perceptions of uncertainty in choosing options and has been demonstrated to be valid and responsive to change. The decisional conflict scale is a 16-item 5-response instrument that reports a score from 0 - 100 with higher scores indicating more conflict (items are summed, divided by 16 and multiplied by 25).

CONTACTS AND LOCATIONS:
Overall Officials: Toni Zhong, MD, MHS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Causarano N, Platt J, Baxter NN, Bagher S, Jones JM, Metcalfe KA, Hofer SO, O'Neill AC, Cheng T, Starenkyj E, Zhong T. Pre-consultation educational group intervention to improve shared decision-making for postmastectomy breast reconstruction: a pilot randomized controlled trial. Support Care Cancer. 2015 May;23(5):1365-75. doi: 10.1007/s00520-014-2479-6. Epub 2014 Oct 29. PMID 25351455
- See also: E-publication link — http://rd.springer.com/article/10.1007%2Fs00520-014-2479-6